CLINICAL TRIAL: NCT00290563
Title: A Multicenter, Double-Blind, Randomized, Placebo- and Active-Controlled, Parallel-Group, Dose-Ranging Study of MK0594 in Patients With Overactive Bladder
Brief Title: Safety and Efficacy of MK0594 to Treat Overactive Bladder (0594-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0594-003; MK0594-003; 2005_102
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: MK0594

SUMMARY:
This study is designed to investigate whether a new drug may offer safe and effective treatment for patients with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with predominantly urge incontinence overactive bladder episodes
* Patients must meet minimum eligibility requirements (e.g., average number of micturitions/day) based on screening diary cards

Exclusion Criteria:

* History of Diabetes insipidus, uncontrolled hyperglycemia or hypercalcemia
* Lower urinary tract symptoms associated with benign prostatic hypertrophy
* Active or current Urinary Tract Infections (UTIs)
* Surgery to correct prolapsed uterus or stress incontinence

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2006-02-21 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-09-24 (Actual)

PRIMARY OUTCOMES:
Change in baseline in average daily micturitions as recorded on patient voiding diaries. | Duration of Trial
  Change in baseline in average daily micturitions as recorded on patient voiding diaries.

SECONDARY OUTCOMES:
The incidence of dry mouth. | Duration of Treatment
  The incidence of dry mouth.
Average daily strong urgency, total incontinence, and Urge UI episodes from voiding diaries. | Duration of Treatment
  Average daily strong urgency, total incontinence, and Urge UI episodes from voiding diaries.
Global assessment of improvement in UI, perception of urgency, and bother of UI symptoms. | Duration of Treatment
  Global assessment of improvement in UI, perception of urgency, and bother of UI

REFERENCES:
- [Derived] Frenkl TL, Zhu H, Reiss T, Seltzer O, Rosenberg E, Green S. A multicenter, double-blind, randomized, placebo controlled trial of a neurokinin-1 receptor antagonist for overactive bladder. J Urol. 2010 Aug;184(2):616-22. doi: 10.1016/j.juro.2010.03.147. Epub 2010 Jun 19. PMID 20639026